CLINICAL TRIAL: NCT04953858
Title: Social Network Strategy to Promote HIV Testing and Linkage to HIV Services Among Young Men Who Have Sex With Men and Transgender Women in Thailand
Brief Title: SNS to Increase HIV Testing Uptake and Linkage to Double Cascade Services Among Adolescent MSM and TGW in Thailand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SNS project
Record Dates: First submitted 2021-05-04; First posted 2021-07-08 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2021-04

CONDITIONS: Social Network Strategy; HIV Self Testing; Men Who Have Sex With Men
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Intervention Model Description: Potential recruiters will be approached in routine adolescent HIV treatment and services and those enrolled will approach peers to become network members who then come in for HIV testing
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Social Network Strategy (Other): All study participants will receive social network strategy intervention as linkage method to receive HIV testing and care
  Interventions: Other: Social network strategy (SNS)

INTERVENTIONS:
Other: Social network strategy (SNS) — SNS utilizes peers to reach and recruit their network members into HIV services, therefore having the advantage that recruiters with different behavioral risks and HIV statuses are likely to have access to a wide variety of HIV at risk populations

SUMMARY:
UNAIDS aims to end AIDS by 2030 using "90-90-90" diagnosis-treatment-viral suppression targets. Thailand has achieved elimination of HIV mother-to-child transmission, but continues to see new infections among adolescent men who have sex with men (YMSM) and transgender women (YTGW). Reaching and engagement of key populations to HIV services remains a major challenge, with differentiated care needed to address this. Investigators propose a study on outreach for HIV at-risk adolescents using peer-led social network strategies (SNS), linkage to facility-based HIV self-testing, and same day HIV prevention or treatment. The study will focus on the 15-19 year age group who have the highest HIV incidence in Thailand (6.9-10 per 100 person years, PY), but will also include young adults aged 20- 24 years of age, due to their frequently intertwining sex networks and very similar HIV incidence of 4.9-7.2 per 100 PY.

Eight hundred adolescent and young adult (AYA) MSM and TGW aged between 15-24 years will be recruited into a double HIV cascade care system. AYA aged between 15-24 years will be trained as recruiters to approach and refer their peers, 'network members' (NMs) to our adolescent clinic. NMs will be offered a choice of either blood-based or oral fluid-based HIV self-testing. HIV positive cases will be offered same-day antiretroviral therapy (SDART) and high-risk adolescents will be offered same day preexposure prophylaxis (PrEP). The project will be conducted at adolescent differentiated care services previously established by CIPHER grants in Thailand, located at King Chulalongkorn Memorial Hospital (KCMH), Bangkok. It will inform both Thailand and other Asia-Pacific region countries with similar epidemic patterns through an implementation research lens on strategies to engage YMSM and YTGW into HIV services, which investigators believe will make high-impact contributions to our collective ultimate goal of ending AIDS.

ELIGIBILITY:
Recruiters

Inclusion Criteria:

* ages 15-24 years
* assigned male gender at birth
* self-defined gender identity of either MSM or TGW
* any one of the following: living with HIV, using HIV pre-exposure prophylaxis, receiving intermittent HIV testing for ongoing HIV risk
* good rapport with King Chulalongkorn Memorial Hospital (KCMH) Adolescent Health Clinic, knowledgable on HIV and comfortable discussing HIV with peers

Network Members

Inclusion Criteria:

* ages 15-24 years
* assigned male gender at birth
* self-defined gender identity of either MSM or TGW
* self-reported oral and/or anal sex with a man in the past 12 months and at risk of HIV infection (multiple sex partners in the preceding 6 months and/or inconsistent condom use)
* no history of HIV testing or last HIV test > 3 months prior to study entry

Exclusion Criteria:

* Known to be living with HIV

Ages: 15 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Men who have sex with men (MSM) or transgender women (TGW)
Enrollment: 202 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
The effectiveness of using social network strategies to increase HIV testing uptake in YMSM and YTGW. | 24 months
  Effectiveness will be measured by proportion of first-time testers among participants enrolled, defined as number of first-time testers divided by total number enrolled. SNS strategies are considered effective when proportions exceed 50 percent. Descriptive statistics of first-time tester characteristics, HIV risk factors, and their recruiter's characteristics will be described.

SECONDARY OUTCOMES:
Pre-exposure prophylaxis (PrEP) uptake among HIV negative at-risk adolescents | 24 months
  PrEP uptake is defined as the number of participants agreeing to initiate PrEP divided by the total number of HIV negative participants enrolled and association of PrEP uptake with factors include recruiter's characteristics will be evaluated utilizing logistic regression to calculate odd ratios and 95 percent confident intervals.
Viral suppression at 6 months for those initiated on antiretroviral treatment among newly diagnosed HIV positive adolescents | 24 months
  Proportions of viral suppression seen at 6 months for those initiated on antiretroviral treatment among newly diagnosed HIV positive adolescents will be calculated. Descriptive statistics will used to describe this group of the sample. Comparison of characteristics between those viral suppressed and not virally suppressed will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- The Division of Infectious Diseases, Department of Pediatrics, Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand